CLINICAL TRIAL: NCT01901458
Title: Prospective Randomized Trial Comparing Efficiency of Peripheral Blood Progenitor Cell Collection in Allogeneic Donors Using the Spectra Optia® IDL Set in Comparison With the Spectra Optia® MNC Collection Set
Brief Title: Two Different Collection Sets for Peripheral Blood Progenitor Cell Apheresis With Spectra Optia®
Acronym: optiMaL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Terumo BCT (Industry); Chugai Pharma USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITZ-003; CIV-13-10-011663 (Other: EUDAMED)
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Allogeneic Donors; Granulocyte Colony-stimulating Factor (G-CSF) Mobilized
Keywords: apheresis; peripheral blood progenitor cells; peripheral blood stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDL-Set (Experimental): Peripheral blood progenitor cell apheresis in G-CSF mobilized allogeneic donors using the Spectra Optia® IDL-Set in combination with the Spectra Optia® cell separator and the WBC-D program
  Interventions: Device: Spectra Optia® IDL-Set
- MNC-Set (Active Comparator): Peripheral blood progenitor cell apheresis in G-CSF mobilized allogeneic donors using the Spectra Optia® Collection Set in combination with the Spectra Optia® cell separator and the MNC program
  Interventions: Device: Spectra Optia® Collection Set

INTERVENTIONS:
Device: Spectra Optia® IDL-Set — Peripheral blood progenitor cell apheresis in G-CSF mobilized allogeneic donors using the Spectra Optia® cell separator
  Arms: IDL-Set
Device: Spectra Optia® Collection Set — Peripheral blood progenitor cell apheresis in G-CSF mobilized allogeneic donors using the Spectra Optia® cell separator
  Arms: MNC-Set

SUMMARY:
The study will determine the advantage of the Spectra Optia® IDL set compared to the standard collection set for collection of peripheral blood progenitor cells using the Spectra Optia® apheresis system. The study will assess the reduction of apheresis time to obtain the required amount of hematopoietic progenitor cells.

DETAILED DESCRIPTION:
Peripheral blood progenitor cells (PBPC) collected by apheresis are the most common stem cell source for allogeneic hematopoietic stem cell transplantation.

Recently, Terumo BCT introduced a novel automated apheresis system for PBPC collection. The Spectra Optia® apheresis system uses the Spectra Optia® Collection set and the MNC software for PBPC collection. This system combines continuous centrifugation (high g) and subsequent cellular collection into an elutriation chamber, where the platelets are elutriated from mononuclear cells. An optical sensor detects when red blood cells begin to be elutriated and subsequently triggers the collection of the buffy coat into the product bag by flushing the chamber with donor plasma. Thus PBPCs are harvested intermittently. In contrast, the same apheresis systems in combination with the Spectra Optia® IDL set and the WBC-D software, which has been designed to perform leukodepletion procedures, permits continuous PBPC centrifugation (low g) and harvesting.

The investigators hypothesis is that the use of the IDL set with manual adaption of the WBC-D-software allows a more efficient PBPC collection compared to the collection set which is recommended for PBPC collection. The apheresis time to collect the same amount of target cells dependent on the donors peripheral blood count will be shortened. In addition, the investigators want to compare both systems with respect to the cellular composition of the apheresis product and the donors platelet loss and coagulation parameters during apheresis.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent to participate in the study
* meets german eligibility criteria (ZKRD-Standards, hemotherapy guidelines) for peripheral blood stem cell donation
* has been treated with G-CSF 10 µg per kg per day for 5 days

Exclusion Criteria:

* demand of concurrent plasma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Throughput (TP) | Day 1
  Efficiency of peripheral blood progenitor cell collection measured as throughput (collection rate (CR) per minute)

SECONDARY OUTCOMES:
CR per total blood volume (TBV) | Day 1
  Efficiency of peripheral blood progenitor cell collection measured as CR per TBV
Collection efficiency (CE) 1 | Day 1
  Percentage of harvested cells per processed cells (calculated by use of the peripheral blood progenitor cell counts pre and post apheresis)
CE2 | Day 1
  Percentage of harvested cells per processed cells (calculated by use of the peripheral blood progenitor cell count pre apheresis)
Product T cells | Day 1
  % T cells as a definition of the cellular composition of the product
Product NK cells | Day 1
  % NK cells as a definition of the cellular composition of the product

OTHER OUTCOMES:
levels of electrolytes before and after apheresis | day 1, day 30
  sodium, potassium and calcium are measured before and after apherese and 30 days after collection
kinetics of peripheral blood cell count | day 1, day30
  measurement of the peripheral blood cell count before and after apheresis and 30 days after collection
Peripheral blood CD62P before and after apheresis | day 1
  Percentage of CD62P positive platelets as a measure of platelet activation during apheresis

CONTACTS AND LOCATIONS:
Overall Officials: Johannes C Fischer, MD, Principal Investigator — Heinrich Heine University Hospital Duesseldorf
Locations (2):
- Germany (2):
  - Cellex GmbH / Zentrum für Zellgewinnung (Standort Köln), Cologne
  - Institut für Transplantantionsdiagnostik und Zelltherapeutika, Düsseldorf